CLINICAL TRIAL: NCT06600204
Title: Comparison of SPECT/CT Perfusion and Volumetric CT Volume to Predict Postoperative Pulmonary Function After Segmentectomy
Brief Title: Comparison of SPECT/CT Perfusion and Volumetric CT Volume
Acronym: VOLSEP
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI070; Retrospective study (Other: CHRU of NANCY)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent a single or multiple segmentectomy: Patients who underwent a single or multiple segmentectomy in the thoracic surgery department of the Nancy University Hospital between April 2021 and July 2023
  Interventions: Other: lung scintigraphy

INTERVENTIONS:
Other: lung scintigraphy — Use the SPECT/CT to predict pulmonary function

SUMMARY:
The main aim of this study is to show that single photon emission tomography/Computer tomography (SPECT/CT) is a reliable examination to predict postoperative pulmonary function after segmentectomy, by comparing this predicted function to that measured at 1 and 6 months.

DETAILED DESCRIPTION:
Lung cancer has a high prevalence, incidence and mortality in France and worldwide. Surgical treatment, possible only at an early stage, improves the prognosis of patients. In addition, the increasing accessibility of chest CT scans allows early detection and monitoring of small pulmonary nodules. As a result, more conservative surgical techniques are becoming increasingly important, including segmentectomy.

Among patients for whom it is indicated, the preoperative assessment involves the evaluation of pulmonary function and the prediction of postoperative pulmonary function in order to validate the feasibility of surgery. To do this, several methods have been described: anatomical methods (segment counting), radiological imaging methods (CT, DECT, perfusion MRI), and nuclear imaging methods (planar perfusion and/or ventilation pulmonary scintigraphy, SPECT pulmonary perfusion scintigraphy), some of which are hybrid (SPECT/CT). The use of SPECT/CT to predict postoperative pulmonary function is routinely practiced, and its reliability, accuracy, and concordance with measured postoperative pulmonary function are well demonstrated for pneumectomy and lobectomy. For more conservative surgeries, the data in the literature remain uncertain. However, being able to predict pulmonary function is essential, both to justify the feasibility of the intervention, but also to target the most fragile patients and intensify their postoperative respiratory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Person having received full information on the organization of the research and not having opposed the exploitation of this data
* Patients having benefited from a single or multiple segmentectomy within the thoracic surgery department of the CHRU of Nancy during the period April 2021 to June 2023
* Patients having a complete pre-operative assessment (SPECT/CT, volumetric CT and EFR)
* Patients having 2 post-operative assessments (respiratory functional exploration (EFR) at approximately 1 month post-operatively and 6 months post-operatively).

Exclusion Criteria:

* Patients who underwent more extensive surgery (lobectomy, pneumectomy) or less extensive surgery (wedge).
* Patient who did not have a complete preoperative assessment (SPECT/CT or volumetric CT or missing respiratory functional exploration EFR).
* Patient who did not have a complete postoperative assessment (missing respiratory functional exploration EFR at 6 months).

NB: the absence of respiratory functional exploration EFR at 1 month postoperatively is not an exclusion criterion

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study including patients who underwent preoperative SPECT/CT pulmonary perfusion scintigraphy examination in the nuclear medicine department, from April 2021 to June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate that SPECT/CT is a reliable examination for predicting postoperative pulmonary function after segmentectomy, by comparing this predicted function to that measured at 1 and 6 months. | 7 months
  Predicted postoperative pulmonary function using SPECT/CT (% perfusion participation of the removed segment(s)).
  Postoperative pulmonary function measured at 1 month Postoperative pulmonary function measured at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of NANCY, Vandœuvre-lès-Nancy, France